CLINICAL TRIAL: NCT06946888
Title: Effects of Acupressure on Nurses' Psychological Distress, Anxiety, Depression, Job Stress, Occupational Burnout, and Resilience
Brief Title: Effects of Acupressure on Nurses' Psychological Distress, Depression, Job Stress, Occupational Burnout, and Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Li-Ying Lin, Nursing Supervisor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KSVGH24-CT6-13
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Results first posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Psychological Distress; Anxiety; Depression; Nurses; Acupressure
Keywords: Nurses; Acupressure; Occupational stress; Burnout, professional; Resilience, psychological; Anxiety; Depression; Psychological distress
MeSH Terms: conditions — Anxiety Disorders; Depression; Occupational Stress; Burnout, Professional | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, single-blind, parallel-controlled trial. Eligible clinical nurses will be randomly assigned (1:1) to an intervention group or a control group. The intervention group will receive self-acupressure instructions on Shenmen and Neiguan points twice a day for two weeks, and record each treatment process. The control group will continue to use their usual stress and emotional distress coping strategies without any intervention. Both groups will be required to complete a validated questionnaire covering emotional distress, mood, anxiety, depression, stress, fatigue and resilience. Assessments will be conducted weekly for two months (including pre-test (baseline week 0) and follow-up for two months (weeks 1-8), a total of 9 times) to evaluate the effectiveness of self-acupressure compared with usual care.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Care continued in the original manner without any intervention.
- Intervention group (Acupressure) (Experimental): Participants perform self-acupressure on the Shenmen and Neiguan points twice daily for 2 weeks.
  Interventions: Behavioral: Acupressure

INTERVENTIONS:
Behavioral: Acupressure — Participants in this group will receive instruction on how to perform self-acupressure targeting two specific acupoints on the hands: Shenmen and Neiguan. The acupressure protocol includes pressing each acupoint approximately 15 times (about 30 seconds), with a total of four acupoints per session (both hands), for approximately 2 minutes per session. Pressure should be applied until a sensation of soreness, numbness, fullness, or slight pain is felt (equivalent to about 3 kg of pressure). Participants are asked to perform self-acupressure twice daily (once in the afternoon and once before bedtime, adjustable based on personal schedule) for a total of 2 weeks. They will record their practice using a daily log and continue to complete psychological and emotional outcome questionnaires weekly over a 2-month follow-up period.
  Arms: Intervention group (Acupressure)

SUMMARY:
This measurement aims to understand the effect of self-acupressure on the Shenmen Point (神門) and (內關) points on the hand on emotional distress, anxiety, depression, stress, work fatigue and adaptability of clinical nurses. The main questions it aims to answer are:

Whether acupressure can reduce emotional distress, anxiety, depression, stress and work fatigue in nursing staff.

Participants will:

1. Enforcement measures:

1. Acupressure group: Perform self-acupressure twice a day, each time for about 2 minutes, and record the acupressure records every day for 2 consecutive weeks.
2. Original method group: followed the original self-coping method. 2. After the intervention began, participants completed study questionnaires weekly for two months.

DETAILED DESCRIPTION:
1. Purpose of the Study:

   The goal of this study is to understand emotional distress, anxiety, depression, stress, workplace fatigue, and resilience among clinical nurses, as well as the factors related to these conditions. Investigators also want to evaluate the effects of different coping methods-either by self-pressing specific acupuncture points (Shenmen and Neiguan on the hand) or using usual ways of managing stress and anxiety.
2. About the Acupressure Points:

   • Shenmen Point (神門): Shenmen, located on the inner wrist, is a key point on the Heart Meridian. It's often used in traditional Chinese medicine to calm the mind, ease anxiety, help with sleep problems, headaches, and emotional fatigue.

   • Neiguan Point (內關): Neiguan is located on the inner forearm. Pressing this point can help relieve stress, reduce bloating, calm palpitations, and improve sleep. It's often used when feeling tense or anxious.

   • Usual Coping Methods: If participants are assigned to this group, participants will simply continue handling stress and anxiety the way you normally do.
3. Who Can Join the Study:

   Participants can join this study if:
   * A clinical nurse aged 20 or older.
   * Participants screening results show a distress score of 3 or above, or a mood thermometer score of 4 or above.
   * Participants are willing and able to fill out questionnaires at specific times over the next two months.

   Participants cannot join this study if:
   * Participated in a similar study within the last month.
   * Currently work in administrative or non-patient care units (like the supply center).
   * Are currently pregnant.
4. Study Procedures:

   If participants agree to participate and sign the consent form, researchers will ask participants to fill out several questionnaires. These will cover basic info, emotional distress, mood, depression, anxiety, work stress, fatigue, and resilience. It takes about 10-20 minutes to complete.

   If participants distress score is 3 or higher, or your mood score is 4 or higher, participants will be randomly assigned to one of two groups:

   • Acupressure Group: Participants will learn how to press the Shenmen and Neiguan acupoints on their hands and press them twice a day (about 2 minutes each time) for 2 weeks. participants will also keep a simple daily log of your acupressure practice.

   • Usual Care Group: Participants will continue with usual ways of coping and fill out a short daily emotional self-assessment form.

   Investigators will check in with participants every week using the same set of questionnaires to track changes for two months. In total, participants will be asked to fill out the survey 9 times.
5. Possible Side Effects and How to Handle Them:

   • From the Acupressure: When pressing the Shenmen or Neiguan points, participants might feel a sensation like soreness, tingling, pressure, or slight pain-this is normal and usually tolerable. There's no research showing any harmful side effects from pressing these points. If it ever feels too uncomfortable, participants can adjust the pressure.

   • From Participation: The risks of participating in this study were similar to participants' normal, everyday experiences. Participants were free to stop at any time if they felt sick or uncomfortable during the study. Participants can also contact the program's emergency contacts.
6. Expected Benefits:

   Past research and traditional practice have shown that pressing the Shenmen and Neiguan points can help reduce anxiety, stress, insomnia, and related symptoms. While the researchers cannot guarantee that this study will help individual participants, it may help healthcare professionals understand ways to better support caregivers and could benefit others in the future.
7. The researcher's requirements for participants during the study:

   * Please do not participate in other similar clinical studies while participating in this clinical study.
   * Please fill in the daily log on time and truthfully.
   * Provide accurate information in the questionnaire.
8. Participants' privacy is protected:

Researchers will only collect information necessary for this study. All personal data and survey responses of participants will remain confidential. The researcher will not use the participant's name or personal identification, but will assign a code to the participant so that the participant's identity remains anonymous in all records.

ELIGIBILITY:
Inclusion Criteria:

* Clinical nurses aged 20 years or older from a designated medical center.
* Nurses who score ≥3 on the emotional distress thermometer or ≥4 on the Brief Symptom Rating Scale (BSRS-5) based on self-reported questionnaires.
* Able and willing to complete the required study questionnaires during the 2-month study period.

Exclusion Criteria:

* Nurses who refuse to participate after being informed about the study or are unable to comply with the study protocol.
* Nurses working in non-patient-care units (e.g., administrative departments or supply centers).
* Pregnant nurses.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ying Lin, PhD, Principal Investigator — supervise
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Zuoying District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou XQ, Han YF, Xu MX. Effects of different intervention methods on psychological anxiety, stress, and fatigue among healthcare workers during COVID-19 pandemic: a systematic review and meta-analysis. Eur Rev Med Pharmacol Sci. 2024 Feb;28(4):1614-1623. doi: 10.26355/eurrev_202402_35491. PMID 38436194
- [Background] Yang X, Liu Q, Wu X. Meta-Analysis of the Clinical Efficacy of Auricular Acupressure on Patients with Depression. Alpha Psychiatry. 2025 Feb 28;26(1):38776. doi: 10.31083/AP38776. eCollection 2025 Feb. PMID 40110387
- [Background] Wu X, Tu M, Yu Z, Cao Z, Qu S, Chen N, Jin J, Xiong S, Yang J, Pei S, Xu M, Wang J, Shi Y, Gao L, Xie J, Li X, Fang J, Shao X. The efficacy and cerebral mechanism of intradermal acupuncture for major depressive disorder: a multicenter randomized controlled trial. Neuropsychopharmacology. 2025 Jun;50(7):1075-1083. doi: 10.1038/s41386-024-02036-5. Epub 2024 Dec 8. PMID 39648209
- [Background] Peng Z, Zheng Y, Yang Z, Zhang H, Li Z, Xu M, Cui S, Lin R. Acupressure: a possible therapeutic strategy for anxiety related to COVID-19: a meta-analysis of randomized controlled trials. Front Med (Lausanne). 2024 Mar 21;11:1341072. doi: 10.3389/fmed.2024.1341072. eCollection 2024. PMID 38576710
- [Background] Pachi A, Sikaras C, Melas D, Alikanioti S, Soultanis N, Ivanidou M, Ilias I, Tselebis A. Stress, Anxiety and Depressive Symptoms, Burnout and Insomnia Among Greek Nurses One Year After the End of the Pandemic: A Moderated Chain Mediation Model. J Clin Med. 2025 Feb 10;14(4):1145. doi: 10.3390/jcm14041145. PMID 40004676
- [Background] Li J, Zhang K, Zhao T, Huang W, Hou R, Wang S, Zhao M, Guo Y. Acupressure for depression: A systematic review and meta-analysis. Asian J Psychiatr. 2024 Feb;92:103884. doi: 10.1016/j.ajp.2023.103884. Epub 2023 Dec 23. PMID 38171225
- [Background] Hong WK, Kim YJ, Lee YR, Jeong HI, Kim KH, Ko SG. Effectiveness of electroacupuncture on anxiety: a systematic review and meta-analysis of randomized controlled trials. Front Psychol. 2023 Dec 19;14:1196177. doi: 10.3389/fpsyg.2023.1196177. eCollection 2023. PMID 38173848
- [Background] Elliott D. Comparison of three instruments for measuring patient anxiety in a coronary care unit. Intensive Crit Care Nurs. 1993 Sep;9(3):195-200. doi: 10.1016/0964-3397(93)90027-u. PMID 8400749
- [Background] Donovan KA, Grassi L, McGinty HL, Jacobsen PB. Validation of the distress thermometer worldwide: state of the science. Psychooncology. 2014 Mar;23(3):241-50. doi: 10.1002/pon.3430. Epub 2013 Nov 11. PMID 25160838
- [Background] Dincer B, Inangil D. The effect of Emotional Freedom Techniques on nurses' stress, anxiety, and burnout levels during the COVID-19 pandemic: A randomized controlled trial. Explore (NY). 2021 Mar-Apr;17(2):109-114. doi: 10.1016/j.explore.2020.11.012. Epub 2020 Dec 3. PMID 33293201
- [Background] Bal SK, Gun M. The effects of acupressure on pain, anxiety and vital signs in patients undergoing coronary angiography: A randomized and sham-controlled trial. Explore (NY). 2024 Jan-Feb;20(1):101-109. doi: 10.1016/j.explore.2023.07.001. Epub 2023 Jul 4. PMID 37429762
- [Background] Amiri S, Mahmood N, Javaid SF, Khan MA. The Effect of Lifestyle Interventions on Anxiety, Depression and Stress: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. Healthcare (Basel). 2024 Nov 13;12(22):2263. doi: 10.3390/healthcare12222263. PMID 39595461
- [Background] Alghamdi R, Bahari G. Shift Work, Psychological Health Disorders, and Job Security Among Nurses: A Cross-Sectional Study. Healthcare (Basel). 2025 Jan 22;13(3):221. doi: 10.3390/healthcare13030221. PMID 39942410
- [Background] Turkili S, Karaman A, Cam Yanik T, Altun Ugras G, Yuksel S, Turkili S, Tasdelen B. The Effects of Acupressure on Preoperative Anxiety, Postoperative Pain, and Nausea and Vomiting in Otolaryngology Patients. J Perianesth Nurs. 2025 Apr;40(2):385-392. doi: 10.1016/j.jopan.2024.05.027. Epub 2024 Sep 19. PMID 39297814
- [Result] Zeiher W, Sego E, Trimmer D, Bowers C. Posttraumatic Stress Disorder in Nurses During a Pandemic: Implications for Nurse Leaders. J Nurs Adm. 2022 Feb 1;52(2):E3-E8. doi: 10.1097/NNA.0000000000001112. PMID 35060955
- [Result] Lin J, Chen T, He J, Chung RC, Ma H, Tsang H. Impacts of acupressure treatment on depression: A systematic review and meta-analysis. World J Psychiatry. 2022 Jan 19;12(1):169-186. doi: 10.5498/wjp.v12.i1.169. eCollection 2022 Jan 19. PMID 35111587
- [Result] Liang R, Tang L, Li L, Zhao N, Yu X, Li J, Wang Q, Cun H, Gao X, Yang W. The effect of pressing needle therapy on depression, anxiety, and sleep for patients in convalescence from COVID-19. Front Neurol. 2024 Dec 18;15:1481557. doi: 10.3389/fneur.2024.1481557. eCollection 2024. PMID 39744118
- [Result] Lee JI, Lee MB, Liao SC, Chang CM, Sung SC, Chiang HC, Tai CW. Prevalence of suicidal ideation and associated risk factors in the general population. J Formos Med Assoc. 2010 Feb;109(2):138-47. doi: 10.1016/S0929-6646(10)60034-4. PMID 20206838
- [Result] Katsiroumpa A, Moisoglou I, Papathanasiou IV, Malliarou M, Sarafis P, Gallos P, Konstantakopoulou O, Rizos F, Galanis P. Resilience and Social Support Protect Nurses from Anxiety and Depressive Symptoms: Evidence from a Cross-Sectional Study in the Post-COVID-19 Era. Healthcare (Basel). 2025 Mar 7;13(6):582. doi: 10.3390/healthcare13060582. PMID 40150432
- See also: Effects and safety of auricular acupressure on depression and anxiety in isolated COVID-19 patients: A single-blind randomized controlled trial. — https://www.frontiersin.org/journals/psychiatry/articles/10.3389/fpsyt.2022.1041829/full
- See also: A survey on the current status of resilience among healthcare professionals and the development of a resilience scale: A sample from a hospital in southern Taiwan. — https://doi.org/10.6174/JHM.201912_20(4).325
- See also: Epidemiological survey of depressive disorder in Kaohsiung Metropolis: Development of a culture-relevant Taiwanese Depression Screening Questionnaire. — https://doi.org/10.6141/TW-SRDA-E88067-1
- See also: Using the BSRS-5 to predict suicidal ideation among community residents. — https://doi.org/10.30126/NSPN.201003.0003
- See also: Development and validation of the Chinese version of the Copenhagen Burnout Inventory. — https://doi.org/10.6288/TJPH2008-27-05-01

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical nurses aged ≥20 years were pre-screened with a questionnaire, and those with an emotional distress score ≥3 (0-10 points) or an emotional thermometer score ≥4 after screening were included (this was the week 0 of enrollment).
Pre-assignment Details: Among those who met the criteria of emotional distress score ≥ 3 points (0-10 points) or emotional thermometer score ≥ 4 points, 160 subjects were selected and randomly divided into a control group or an acupoint massage group for an 8-week follow-up (the acupoint massage group was required to press the Shenmen and Neiguan acupoints on their own in the first two weeks, and the control group received no intervention measures), and filled out questionnaires every week for post-test follow-up.
Period: Overall Study
Arm/Group | Control Group | Intervention Group (Acupressure)
Started | 80 | 80
Completed | 80 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A pretest was conducted on clinical nurses in medical centers aged ≥20 years, and 160 nurses with emotional distress ≥3 points or emotional thermometer ≥4 points were selected as intervention subjects. A randomized controlled trial was conducted, in which nurses were randomly assigned to the intervention group and the control group by computer random numbering, and an eight-week follow-up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group (Acupressure) | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] — The age of 160 subjects was analyzed by MEAN and Standard Deviation Population: After collecting the data of 160 subjects, we will analyze them into MEAN and Standard Deviation to see the overall distribution.
  years | 34.45 (12.04) | 30.44 (10.03) | 32.59 (11.281)
Sex: Female, Male [Count of Participants; unit: Participants] — 160 subjects filled in the proportion of each group according to gender Population: Use percentages to look at the distribution of male and female students in the control and intervention groups.
  Participants
    Female | 77 | 74 | 151
    Male | 3 | 6 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — The 160 subjects were mainly clinical nurses at Kaohsiung Veterans General Hospital in Taiwan. Population: All 160 subjects were admitted in Taiwan, so the number of people can be used to represent it.
  Participants
    Taiwan | 80 | 80 | 160

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms
Description: Depressive symptoms were assessed using the Taiwanese Depression Scale, which has demonstrated strong psychometric properties in Taiwanese populations. The TDS consists of 18 items rated on a 4-point Likert scale: 0 = none or seldom (less than one day per week), 1 = sometimes (one to two days per week), 2 = often (three to four days per week), and 3 = almost always (five to seven days per week). Total scores range from 0 to 54, with higher scores indicating greater severity of depressive symptoms.
  The results from Lee et al. (2000) demonstrated that the TDS had excellent reliability and validity. The Cronbach's alpha coefficient was 0.90, and the area under the receiver operating characteristic (ROC) curve was 0.92. The TDS also showed good concurrent validity, with a sensitivity of 0.89 and specificity of 0.92 at a cutoff score of 19.
  In the present study, the TDS demonstrated excellent internal consistency, with a Cronbach's alpha of .94.
Time Frame: At baseline(weeks 0) and once weekly for 8 weeks(weeks 1-8)
Population: After the pre-test questionnaire assessment (baseline week 0), the subjects (control group/intervention group) will be followed up with a weekly questionnaire survey for eight weeks (weeks 1 to 8) after the start of the program. The depression questionnaire will obtain data for a total of nine weeks (baseline week 0 and follow-up weeks 1 to 8) and conduct data analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Group: Care continued in the original manner without any intervention.Participants were asked to fill out a questionnaire (including the Taiwanese Depression Scale) every week (starting day + 7 days/14 days/21 days/28 days, etc.) for 2 months after the start of the program. The results were analyzed after the 2-month follow-up.
- Intervention Group (Acupressure): Participants performed self-acupressure on the Shenmen and Neiguan acupoints twice a day for two weeks. Participants were asked to fill out a questionnaire (including the Taiwanese Depression Scale) every week (starting day + 7 days/14 days/21 days/28 days, etc.) for 2 months after the start of the program. The results were analyzed after the 2-month follow-up.
Arm/Group | Control Group | Intervention Group (Acupressure)
Number analyzed (Participants) | 80 | 80
score on a scale
  Tracking Week 1 | 11.76 (7.20) | 11.55 (6.76)
  Tracking Week 2 | 11.70 (7.51) | 10.84 (8.12)
  Tracking Week 3 | 12.05 (8.22) | 10.86 (7.51)
  Tracking Week 4 | 13.35 (8.39) | 10.59 (9.02)
  Tracking Week 5 | 12.54 (8.84) | 10.95 (8.98)
  Tracking Week 6 | 12.66 (9.63) | 10.93 (9.22)
  Tracking Week 7 | 12.05 (9.24) | 10.16 (8.19)
  Tracking Week 8 | 12.31 (10.64) | 10.51 (8.62)
  Tracking Week 0 | 13.03 (7.37) | 13.00 (7.33)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group (Acupressure); Generalized estimating equations (GEE) were chosen over repeated-measures analysis of variance or generalized linear mixed models because they provide estimates of the population mean, are robust to correlated error specifications, can accommodate missing data under the MAR/MCAR assumptions, and do not require sphericity. All tests were two-tailed, with α = 0.05; Test type: Other — A generalized estimating equation (GEE) model included group (intervention group vs. control group), week (categorical: 0-8), group × week interaction, and age as covariates. Robust (sandwich) standard errors were used. Regression coefficients (B), standard errors, Wald chi-squared statistics, 95% confidence intervals, and p-values for group × week comparisons are reported; p = 0.837, Generalized Estimating Equations, GEE — This is the first week of tracking. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 1
Statistical Analysis 2: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.428, Generalized Estimating Equations, GEE — This is the second week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 2
Statistical Analysis 3: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.269, Generalized Estimating Equations, GEE — This is the third week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 3
Statistical Analysis 4: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.015, Generalized Estimating Equations, GEE — This is the fourth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 4
Statistical Analysis 5: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.163, Generalized Estimating Equations, GEE — This is the fifth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 5
Statistical Analysis 6: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.140, Generalized Estimating Equations, GEE — This is the sixth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 6
Statistical Analysis 7: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.079, Generalized Estimating Equations, GEE — This is the seventh week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 7
Statistical Analysis 8: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.151, Generalized Estimating Equations, GEE — This is the eighth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 8

2. Primary Outcome: Psychological Distress
Description: Psychological distress was measured using the Brief Symptom Rating Scale-5 (BSRS-5), a validated screening tool for general psychological distress. The BSRS-5 assesses the subjective severity of the following symptoms: (1) anxiety, (2) depression, (3) hostility, (4) low self-esteem, and (5) insomnia. Each symptom was scored on a 5-point Likert scale, ranging from 0 ("not at all") to 4 ("extremely"), with a total score ranging from 0 to 20 points. Higher scores indicate more severe psychological distress.
  Studies have shown that a total score of 3-4 is the optimal threshold for identifying clinically relevant distress based on receiver operating characteristic (ROC) curve analysis. The BSRS-5 showed high accuracy (AUC = 0.92) and good sensitivity (0.83) and specificity (0.86). Therefore, this study used a BSRS-5 total score ≥4 as one of the inclusion criteria to ensure that participants with at least mild psychological distress were included in the study.
Time Frame: At baseline(weeks 0) and once weekly for 8 weeks(weeks 1-8)
Population: After the pre-test questionnaire assessment (baseline week 0), the subjects (control group/intervention group) will be followed up with weekly questionnaires for eight weeks (weeks 1 to 8) after the start of the program, of which the Mood Thermometer (Brief Symptoms Rating Scale, BSRS-5) questionnaire will obtain data for a total of nine weeks (baseline week 0 and follow-up weeks 1 to 8) and conduct data analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Group: Care continued in the original manner without any intervention.Participants were asked to fill out a questionnaire (including the Brief Symptoms Rating Scale) every week (starting day + 7 days/14 days/21 days/28 days, etc.) for 2 months after the start of the program. The results were analyzed after the 2-month follow-up.
- Intervention Group (Acupressure): Participants performed self-acupressure on the Shenmen and Neiguan acupoints twice a day for two weeks. Participants were asked to fill out a questionnaire (including the Brief Symptoms Rating Scale) every week (starting day + 7 days/14 days/21 days/28 days, etc.) for 2 months after the start of the program. The results were analyzed after the 2-month follow-up.
Arm/Group | Control Group | Intervention Group (Acupressure)
Number analyzed (Participants) | 80 | 80
score on a scale
  Tracking Week 1 | 5.65 (3.42) | 5.54 (3.32)
  Tracking Week 2 | 5.54 (3.12) | 5.31 (3.56)
  Tracking Week 3 | 5.05 (3.03) | 4.6 (3.23)
  Tracking Week 4 | 5.53 (3.67) | 4.66 (3.44)
  Tracking Week 5 | 5.28 (3.81) | 4.81 (3.42)
  Tracking Week 6 | 4.99 (3.80) | 4.48 (3.39)
  Tracking Week 7 | 5.09 (3.85) | 4.55 (3.26)
  Tracking Week 8 | 5.05 (4.15) | 4.40 (3.18)
  Tracking Week 0 | 6.53 (3.36) | 6.41 (3.28)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.63, Generalized Estimating Equations, GEE — This is the first week of tracking. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 1
Statistical Analysis 2: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.608, Generalized Estimating Equations, GEE — This is the second week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 2
Statistical Analysis 3: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.244, Generalized Estimating Equations, GEE — This is the third week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 3
Statistical Analysis 4: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.052, Generalized Estimating Equations, GEE — This is the fourth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 4
Statistical Analysis 5: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.229, Generalized Estimating Equations, GEE — This is the fifth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 5
Statistical Analysis 6: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.184, Generalized Estimating Equations, GEE — This is the sixth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 6
Statistical Analysis 7: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.148, Generalized Estimating Equations, GEE — This is the seventh week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 7
Statistical Analysis 8: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.143, Generalized Estimating Equations, GEE — This is the eighth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 8

3. Secondary Outcome: Resilience
Description: This scale assesses an individual's ability to adapt and recover from stress and adversity. Each item is rated on a 5-point Likert scale, ranging from 1 ("strongly disagree") to 5 ("strongly agree"), with a total score ranging from 10 to 50, with higher scores indicating greater resilience.
  Initial validation studies demonstrated strong psychometric properties, including good model fit in confirmatory factor analysis (GFI = 0.973) and excellent internal consistency (Cronbach's α = .91).
  All instruments used in this study were authorized by their original developers and have been psychometrically validated in previous studies. All scales demonstrated good to excellent internal consistency, with Cronbach's α values ranging from 0.84 to 0.95.
Time Frame: At baseline(weeks 0) and once weekly for 8 weeks(weeks 1-8)
Population: After the pre-test questionnaire assessment (baseline week 0), the subjects (control group/intervention group) will be followed up with weekly questionnaires for eight weeks (weeks 1 to 8) after the start of the program, of which the Resilience questionnaire will obtain data for a total of nine weeks (baseline week 0 and follow-up weeks 1 to 8) and conduct data analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Group: Care continued in the original manner without any intervention.Participants were asked to fill out a questionnaire (including the resilience) every week (starting day + 7 days/14 days/21 days/28 days, etc.) for 2 months after the start of the program. The results were analyzed after the 2-month follow-up.
- Intervention Group (Acupressure): Participants performed self-acupressure on the Shenmen and Neiguan acupoints twice a day for two weeks. Participants were asked to fill out a questionnaire (including the resilience) every week (starting day + 7 days/14 days/21 days/28 days, etc.) for 2 months after the start of the program. The results were analyzed after the 2-month follow-up.
Arm/Group | Control Group | Intervention Group (Acupressure)
Number analyzed (Participants) | 80 | 80
score on a scale
  Tracking Week 1 | 38.64 (4.64) | 39.18 (5.22)
  Tracking Week 2 | 38.83 (5.04) | 39.62 (4.87)
  Tracking Week 3 | 38.86 (5.08) | 39.63 (4.81)
  Tracking Week 4 | 39.40 (4.65) | 40.15 (5.64)
  Tracking Week 5 | 39.30 (4.55) | 40.21 (5.49)
  Tracking Week 6 | 39.09 (5.60) | 40.19 (5.38)
  Tracking Week 7 | 39.16 (5.36) | 40.24 (5.48)
  Tracking Week 8 | 39.59 (5.24) | 40.33 (5.70)
  Tracking Week 0 | 38.70 (4.84) | 40.00 (4.94)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.333, Generalized Estimating Equations, GEE — This is the first week of tracking. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 1
Statistical Analysis 2: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.273, Generalized Estimating Equations, GEE — This is the second week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 2
Statistical Analysis 3: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.424, Generalized Estimating Equations, GEE — This is the third week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 3
Statistical Analysis 4: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.482, Generalized Estimating Equations, GEE — This is the fourth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 4
Statistical Analysis 5: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.627, Generalized Estimating Equations, GEE — This is the fifth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 5
Statistical Analysis 6: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.806, Generalized Estimating Equations, GEE — This is the sixth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 6
Statistical Analysis 7: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.786, Generalized Estimating Equations, GEE — This is the seventh week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 7
Statistical Analysis 8: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.497, Generalized Estimating Equations, GEE — This is the eighth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 8

4. Secondary Outcome: Anxiety
Description: Anxiety levels were assessed using the state subscale of the State-Trait Anxiety Inventory (STAI-S). Studies have confirmed the multidimensional factor structure of the Chinese version of the scale and demonstrated good psychometric properties, including adequate convergent and discriminant validity. In this sample, the STAI-S demonstrated excellent internal consistency (Cronbach's α = .95). The STAI-S consists of 20 items that assess anxiety-related feelings, thoughts, and behaviors at the time of assessment. Each item is rated on a 4-point Likert scale ranging from 1 ("not at all") to 4 ("very much"). Items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20 are reverse-scored. The total score ranges from 20 to 80, with scores between 20 and 39 indicating mild anxiety, 40 to 59 indicating moderate anxiety, and 60 to 80 indicating severe anxiety.
Time Frame: At baseline(weeks 0) and once weekly for 8 weeks(weeks 1-8)
Population: After the pre-test questionnaire assessment (baseline week 0), the subjects (control group/intervention group) will be followed up with weekly questionnaires for eight weeks (weeks 1 to 8) after the start of the program. The anxiety questionnaire will obtain data for a total of nine weeks (baseline week 0 and follow-up weeks 1 to 8) and conduct data analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Group: Care continued in the original manner without any intervention.Participants were asked to fill out a questionnaire (including the State Anxiety Scale) every week (starting day + 7 days/14 days/21 days/28 days, etc.) for 2 months after the start of the program. The results were analyzed after the 2-month follow-up.
- Intervention Group (Acupressure): Participants performed self-acupressure on the Shenmen and Neiguan acupoints twice a day for two weeks. Participants were asked to fill out a questionnaire (including the State Anxiety Scale) every week (starting day + 7 days/14 days/21 days/28 days, etc.) for 2 months after the start of the program. The results were analyzed after the 2-month follow-up.
Arm/Group | Control Group | Intervention Group (Acupressure)
Number analyzed (Participants) | 80 | 80
score on a scale
  Tracking Week 1 | 45.18 (10.76) | 44.19 (11.52)
  Tracking Week 2 | 44.64 (10.09) | 43.36 (11.36)
  Tracking Week 3 | 43.93 (10.73) | 41.78 (11.72)
  Tracking Week 4 | 45.00 (10.38) | 42.04 (12.42)
  Tracking Week 5 | 44.58 (10.49) | 42.98 (12.82)
  Tracking Week 6 | 45.01 (11.29) | 42.65 (13.54)
  Tracking Week 7 | 45.49 (11.97) | 44.14 (13.00)
  Tracking Week 8 | 45.18 (13.12) | 41.61 (12.83)
  Tracking Week 0 | 46.15 (9.20) | 45.41 (9.96)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.857, Generalized Estimating Equations, GEE — This is the first week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 1
Statistical Analysis 2: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.684, Generalized Estimating Equations, GEE — This is the second week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 2
Statistical Analysis 3: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.333, Generalized Estimating Equations, GEE — This is the third week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 3
Statistical Analysis 4: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.090, Generalized Estimating Equations, GEE — This is the fourth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 4
Statistical Analysis 5: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.545, Generalized Estimating Equations, GEE — This is the fifth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 5
Statistical Analysis 6: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.251, Generalized Estimating Equations, GEE — This is the sixth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 6
Statistical Analysis 7: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.701, Generalized Estimating Equations, GEE — This is the seventh week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 7
Statistical Analysis 8: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.080, Generalized Estimating Equations, GEE — This is the eighth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 8

5. Secondary Outcome: Job Stress
Description: Perceived job stress was measured using the 14-item Work Pressure Inventory developed by Huang et al. (2017), which has demonstrated good internal consistency. The scale comprises three dimensions: low self-development, workload, and job characteristics. Each item is rated on a 5-point Likert scale ranging from 1 ("strongly disagree") to 5 ("strongly agree"), with total scores ranging from 14 to 70. Higher scores indicate greater perceived occupational stress. In the original validation study, the Cronbach's α coefficients for the three subscales were 0.81, 0.73, and 0.77, respectively. In the present study, the Work Pressure Inventory showed good overall internal consistency (Cronbach's α = .84).
Time Frame: At baseline(weeks 0) and once weekly for 8 weeks(weeks 1-8)
Population: After the pre-test questionnaire assessment (baseline week 0), the subjects (control group/intervention group) will be followed up with weekly questionnaires for eight weeks (weeks 1 to 8) after the start of the program. The Nurse Stress questionnaire will obtain data for a total of nine weeks (baseline week 0 and follow-up weeks 1 to 8) and conduct data analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Group: Care continued in the original manner without any intervention.Participants were asked to fill out a questionnaire (including the Nurse Stress Checklist) every week (starting day + 7 days/14 days/21 days/28 days, etc.) for 2 months after the start of the program. The results were analyzed after the 2-month follow-up.
- Intervention Group (Acupressure): Participants performed self-acupressure on the Shenmen and Neiguan acupoints twice a day for two weeks. Participants were asked to fill out a questionnaire (including the Nurse Stress Checklist) every week (starting day + 7 days/14 days/21 days/28 days, etc.) for 2 months after the start of the program. The results were analyzed after the 2-month follow-up.
Arm/Group | Control Group | Intervention Group (Acupressure)
Number analyzed (Participants) | 80 | 80
score on a scale
  Tracking Week 1 | 45.80 (6.29) | 45.10 (6.87)
  Tracking Week 2 | 45.98 (6.35) | 45.63 (7.14)
  Tracking Week 3 | 45.64 (6.52) | 44.90 (8.33)
  Tracking Week 4 | 45.66 (7.02) | 44.74 (7.71)
  Tracking Week 5 | 45.95 (7.28) | 44.89 (8.08)
  Tracking Week 6 | 45.26 (6.81) | 45.29 (7.58)
  Tracking Week 7 | 45.53 (7.09) | 45.18 (8.30)
  Tracking Week 8 | 45.93 (7.23) | 44.89 (8.11)
  Tracking Week 0 | 45.55 (6.13) | 45.31 (7.79)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.636, Generalized Estimating Equations, GEE — This is the first week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 1
Statistical Analysis 2: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.909, Generalized Estimating Equations, GEE — This is the second week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 2
Statistical Analysis 3: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.627, Generalized Estimating Equations, GEE — This is the third week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 3
Statistical Analysis 4: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.474, Generalized Estimating Equations, GEE — This is the fourth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 4
Statistical Analysis 5: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.378, Generalized Estimating Equations, GEE — This is the fifth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 5
Statistical Analysis 6: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.768, Generalized Estimating Equations, GEE — This is the sixth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 6
Statistical Analysis 7: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.909, Generalized Estimating Equations, GEE — This is the seventh week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 7
Statistical Analysis 8: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.449, Generalized Estimating Equations, GEE — This is the eighth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 8

6. Secondary Outcome: Occupational Burnout
Description: Occupational burnout was assessed using the Chinese version of the Copenhagen Burnout Inventory (CBI), which has demonstrated good psychometric properties in Taiwanese populations. The scale consists of four subscales: personal burnout, work-related burnout, client-related burnout, and overcommitment to work. Each item is rated on a five-point frequency scale: "always" (100), "often" (75), "sometimes" (50), "rarely" (25), and "never" (0). Subscale scores are calculated as the average of the items within each domain, ranging from 0 to 100, with higher scores indicating more severe occupational burnout. The original validation study reported Cronbach's α values above 0.84 across all subscales. In the present study, the scale demonstrated excellent internal consistency (Cronbach's α = .95).
Time Frame: At baseline(weeks 0) and once weekly for 8 weeks(weeks 1-8)
Population: After the pre-test questionnaire assessment (baseline week 0), the subjects (control group/intervention group) will be followed up with weekly questionnaires for eight weeks (weeks 1 to 8) after the start of the program. The workplace fatigue questionnaire will obtain data for a total of nine weeks (baseline week 0 and follow-up weeks 1 to 8) and conduct data analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Group: Care continued in the original manner without any intervention.Participants were asked to fill out a questionnaire (including the occupational burnout) every week (starting day + 7 days/14 days/21 days/28 days, etc.) for 2 months after the start of the program. The results were analyzed after the 2-month follow-up.
- Intervention Group (Acupressure): Participants performed self-acupressure on the Shenmen and Neiguan acupoints twice a day for two weeks. Participants were asked to fill out a questionnaire (including the occupational burnout) every week (starting day + 7 days/14 days/21 days/28 days, etc.) for 2 months after the start of the program. The results were analyzed after the 2-month follow-up.
Arm/Group | Control Group | Intervention Group (Acupressure)
Number analyzed (Participants) | 80 | 80
score on a scale
  Tracking Week 1 | 48.20 (14.77) | 49.05 (15.64)
  Tracking Week 2 | 48.60 (14.92) | 48.44 (17.48)
  Tracking Week 3 | 46.53 (14.19) | 46.46 (17.86)
  Tracking Week 4 | 46.90 (17.19) | 46.86 (17.40)
  Tracking Week 5 | 48.33 (17.21) | 47.43 (17.67)
  Tracking Week 6 | 48.47 (18.48) | 46.62 (17.94)
  Tracking Week 7 | 48.60 (17.46) | 46.53 (19.45)
  Tracking Week 8 | 48.74 (18.80) | 46.24 (19.66)
  Tracking Week 0 | 49.97 (15.19) | 49.79 (15.74)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.593, Generalized Estimating Equations, GEE — This is the first week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 1
Statistical Analysis 2: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.994, Generalized Estimating Equations, GEE — This is the second week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 2
Statistical Analysis 3: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.959, Generalized Estimating Equations, GEE — This is the third week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 3
Statistical Analysis 4: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.946, Generalized Estimating Equations, GEE — This is the fourth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 4
Statistical Analysis 5: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.715, Generalized Estimating Equations, GEE — This is the fifth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 5
Statistical Analysis 6: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.422, Generalized Estimating Equations, GEE — This is the sixth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 6
Statistical Analysis 7: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.379, Generalized Estimating Equations, GEE — This is the seventh week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 7
Statistical Analysis 8: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.302, Generalized Estimating Equations, GEE — This is the eighth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 8

7. Secondary Outcome: Emotional Distress
Description: Emotional distress was measured using the Distress Thermometer (DT), a single self-report screening instrument with a score range of 0 (no distress) to 10 (extreme distress), with higher scores indicating greater emotional distress. The DT demonstrated good psychometric properties in validation studies, with sensitivities ranging from 0.50 to 1.00 (median = 0.83) and specificities ranging from 0.36 to 0.98 (median = 0.68).
  This study used a DT cutoff score of ≥3 as the inclusion criterion. Other studies have shown that the optimal DT cutoff score varies across settings, typically ranging from 3 to 5, while thresholds of ≥4 or ≥5 are commonly used in clinical practice. The use of a score of ≥3 in this study was intended to maximize sensitivity and minimize the risk of underidentifying caregivers considered at high risk for psychological distress.
Time Frame: At baseline(weeks 0) and once weekly for 8 weeks(weeks 1-8)
Population: After the pre-test questionnaire assessment (baseline week 0), the subjects (control group/intervention group) will be followed up with weekly questionnaires for eight weeks (weeks 1 to 8) after the start of the program. A total of nine weeks (baseline week 0 and follow-up weeks 1 to 8) of Distress Thermometer questionnaire data will be obtained and analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Group: Care continued in the original manner without any intervention.Participants were asked to fill out a questionnaire (including the Distress Thermometer) every week (starting day + 7 days/14 days/21 days/28 days, etc.) for 2 months after the start of the program. The results were analyzed after the 2-month follow-up.
- Intervention Group (Acupressure): Participants performed self-acupressure on the Shenmen and Neiguan acupoints twice a day for two weeks. Participants were asked to fill out a questionnaire (including the Distress Thermometer) every week (starting day + 7 days/14 days/21 days/28 days, etc.) for 2 months after the start of the program. The results were analyzed after the 2-month follow-up.
Arm/Group | Control Group | Intervention Group (Acupressure)
Number analyzed (Participants) | 80 | 80
score on a scale
  Tracking Week 1 | 3.95 (1.95) | 3.84 (1.91)
  Tracking Week 2 | 3.59 (1.93) | 3.43 (1.84)
  Tracking Week 3 | 3.41 (1.95) | 3.18 (1.68)
  Tracking Week 4 | 3.48 (2.02) | 3.09 (1.83)
  Tracking Week 5 | 3.35 (1.97) | 3.28 (1.97)
  Tracking Week 6 | 3.38 (1.88) | 3.2 (2.07)
  Tracking Week 7 | 2.93 (1.71) | 3.30 (2.01)
  Tracking Week 8 | 3.26 (1.83) | 3.23 (2.07)
  Tracking Week 0 | 4.01 (1.90) | 3.94 (2.00)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.913, Generalized Estimating Equations, GEE — This is the first week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 1
Statistical Analysis 2: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.802, Generalized Estimating Equations, GEE — This is the second week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 2
Statistical Analysis 3: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.605, Generalized Estimating Equations, GEE — This is the third week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 3
Statistical Analysis 4: Comparison: Control Group vs Intervention Group (Acupressure); Generalized Estimating Equations were used to analyze repeated measures data and to assess the interaction effect between group and time. Potential interfering factors such as age and years of work experience were controlled during the analysis, and the effect size (Cohen's d) and its 95% confidence interval were calculated to assist in interpreting the clinical significance. Statistical analysis was performed using SPSS version XX or R version XX, and the significance level was set at p < 0.05; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.350, Generalized Estimating Equations, GEE — This is the fourth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 4
Statistical Analysis 5: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 1.000, Generalized Estimating Equations, GEE — This is the fifth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 5
Statistical Analysis 6: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.744, Generalized Estimating Equations, GEE — This is the sixth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 6
Statistical Analysis 7: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.202, Generalized Estimating Equations, GEE — This is the seventh week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 7
Statistical Analysis 8: Comparison: Control Group vs Intervention Group (Acupressure); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.918, Generalized Estimating Equations, GEE — This is the eighth week of tracking data. A P value < 0.05 indicated a statistically significant difference; Repeated-measures GEE was used to examine the group × time interaction between week 0 and week 8

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 8 weeks.
Groups:
- Control Group; Intervention Group (Acupressure): From enrollment until end of follow-up, up to 8 weeks.
Arm/Group | Control Group | Intervention Group (Acupressure)
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

LIMITATIONS AND CAVEATS:
1. The data are all self-administered questionnaires, which are affected by recall bias and social expectations.
2. The intervention period is only two weeks, and the intervention period or stimulation frequency can be extended.
3. Other acupoints related to emotional stability are not included, nor are they combined with common auxiliary methods.
4. Multiple workplace factors can be incorporated into the analysis to enhance external validity and reference for practical application.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: The impact of acupressure on nurses in medical center (2024-12-31): https://cdn.clinicaltrials.gov/large-docs/88/NCT06946888/Prot_SAP_000.pdf